CLINICAL TRIAL: NCT00402168
Title: Belatacept Conversion Trial in Renal Transplantation
Brief Title: A Study of BMS-224818 (Belatacept) in Patients Who Have Undergone a Kidney Transplant and Are Currently on Stable Cyclosporine or Tacrolimus Regimen With or Without Corticosteroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-010; LEA29Y
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Abatacept; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Belatacept (Experimental)
  Interventions: Drug: Belatacept
- B: calcineurin inhibitor (CNI)-based immunosuppressive regimen (Active Comparator)
  Interventions: Drug: Cyclosporine A; Drug: Tacrolimus

INTERVENTIONS:
Drug: Belatacept — IV, IV Infusion, 5 mg/kg once every 28 days for one year
  Other Names: BMS-224818
  Arms: A: Belatacept
Drug: Cyclosporine A — Tablets, Oral, Trough of 100-250 ng/mL, 2* daily for one year
  Arms: B: calcineurin inhibitor (CNI)-based immunosuppressive regimen
Drug: Tacrolimus — Tablets, Oral, Trough of 5-10 ng/mL, 2* daily for one year
  Arms: B: calcineurin inhibitor (CNI)-based immunosuppressive regimen

SUMMARY:
The purpose of this study is to learn if conversion to belatacept from cyclosporine or tacrolimus will preserve kidney function in people who have had a kidney transplant. The safety and tolerability of this treatment will also be studied

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women age 18 and older
* 6-36 months after kidney transplant receiving cyclosporine or tacrolimus
* calculated GFR ≥35 and ≤75mL/min/1.73 m²
* subjects must have completed 1 year in the IM103-010ST and remained on study treatment (Long Term Extension)

Key Exclusion Criteria:

* Significant infection
* acute rejection within 3 months
* prior graft loss due to rejection
* pregnancy
* positive crossmatch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (42):
- United States (9):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - National Institute Of Transplantation, Los Angeles, California
  - California Institute Of Renal Research, San Diego, California
  - Ucsf, San Francisco, California
  - University Of Chicago, Chicago, Illinois
  - Pharmacy, First Call Iv, Kenner, Louisiana
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - University Of North Carolina School Of Medicine, Chapel Hill, North Carolina
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (5):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
- Local Institution, Parkville, Victoria, Australia
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Edegem
- Brazil (4):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Bonsucesso, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (4):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Hamilton, Ontario
  - Local Institution, Saskatoon, Saskatchewan
- France (2):
  - Local Institution, Paris, Cedex 15
  - Local Institution, Toulouse
- Germany (2):
  - Charite Berlin Mitte, Berlin
  - Local Institution, Homburg/saar
- India (3):
  - Local Institution, Pāladi, Ahmedabad
  - Local Institution, Nadiād, Gujarat
  - Local Institution, Kochi, Kerala
- Mexico (5):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Df, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, San Luis Potosí City, Snl
  - Local Institution, Tlalpan, C P
- Poland (3):
  - Local Institution, Bydgoszcz
  - Local Institution, Szczecin
  - Local Institution, Warsaw
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Valencia

REFERENCES:
- [Derived] Rostaing L, Massari P, Garcia VD, Mancilla-Urrea E, Nainan G, del Carmen Rial M, Steinberg S, Vincenti F, Shi R, Di Russo G, Thomas D, Grinyo J. Switching from calcineurin inhibitor-based regimens to a belatacept-based regimen in renal transplant recipients: a randomized phase II study. Clin J Am Soc Nephrol. 2011 Feb;6(2):430-9. doi: 10.2215/CJN.05840710. Epub 2010 Nov 4. PMID 21051752
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 173 participants were enrolled, 2 participants discontinued the study following randomization, without receiving any study drug.
Groups:
- Belatacept 5 mg/kg: Belatacept 5 milligrams per kilogram of body weight (mg/kg) given intravenously (IV) every 28 days.
- Calcineurin Inhibitor (CNI): Participants received a calcineurin inhibitor (CNI)-based immunosuppressive regimen, Cyclosporin A (CsA) and tacrolimus (TAC). CsA was to be adjusted to maintain a range of trough serum concentrations of 100 - 250 nanograms per milliliter (ng/mL). TAC doses were to be adjusted to maintain a range of trough serum concentrations of 5 - 10 ng/mL. During the long term (LT) treatment period participants were allowed to switch to belatacept treatment arm. In October 2011 (Year 3), the CNI arm was discontinued. CNI participants were considered to have completed treatment (not discontinued) at that time, if they did not switch to the belatacept arm.
Period: Randomized
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Started | 84 | 89
Completed | 83 | 88
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment (up to 12 Months)
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Started | 83 | 88
Completed | 81 | 86
Not Completed | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — non-specified | 0 | 1
Period: Long Term (LT)
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Started | 81 | 81 (5 completed 12 months, did not enter long term: 1 AE, 1 lack of efficacy, 3 other(non-specified).)
Completed | 70 | 64
Not Completed | 11 | 17
Not completed — Adverse Event | 1 | 5
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 4 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — non-specified | 1 | 2
Period: Switched From CNI to Belatacept in LT
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Started | 38 (Participants switched from CNI to Belatacept during LT period.) | 0 (Out of 81 starting LT period in CNI group, 38 switched from CNI to Belatacept during the LT period.)
Completed | 32 | 0
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 4 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized to a treatment arm.
Groups:
- Belatacept 5 mg/kg: Belatacept 5 mg/kg IV every 28 days.
- Calcineurin Inhibitor (CNI): Participants received a CNI-based immunosuppressive regimen, CsA and TAC. CsA was to be adjusted to maintain a range of trough concentrations of 100 - 250 ng/mL. TAC doses were to be adjusted to maintain a range of trough serum concentrations of 5 - 10 ng/mL. During the LT period, participants were allowed to switch to the belatacept arm. In October 2011 (Year 3), the CNI arm was discontinued. CNI participants were considered to have completed treatment (not discontinued) at that time, if they did not switch to the belatacept arm.
- Total: Total of all reporting groups
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI) | Total
Number analyzed (Participants) | 84 | 89 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.5) | 44.3 (13.0) | 44.8 (13.2)
Age, Customized [Number; unit: participants]
  18 - 45 years | 42 | 47 | 89
  46 - 65 years | 37 | 36 | 73
  Greater than (>) 65 years | 5 | 6 | 11
Gender [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 66 | 60 | 126

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Calculated Glomerular Filtration Rate (GFR) With Imputed Values to 6 Months Post Randomization - All Randomized Participants (Intent-to-Treat Population)
Description: Calculated GFR assessment used the modification of diet in renal disease (MDRD) formula. GFR was measured as mL/min/1.73 m^2. For death or graft loss participants, calculated GFR (cGFR) value 10 was used, for other participants who had a post baseline cGFR value missing, but had baseline value and at least 2 post baseline values available, which were at least 120 days apart, linear regression model was used to impute the cGFR value. Baseline = value at screening.
Time Frame: Baseline to 6 months post randomization
Population: Intent-to-Treat (ITT) population: all randomized participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Groups:
- Belatacept 5 mg/kg: Belatacept 5 mg/kg was given IV every 28 days.
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 82 | 87
mL/min/1.73 m^2 | 6.9 (11.97) | 1.1 (9.84)

2. Secondary Outcome: Number of Participants With Acute Rejection (AR) by Months 6 and 12 Post Randomization - All Randomized Participants
Description: AR defined: if either a or b was satisfied: a: the reason for clinical suspicion was reported to be an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; or an unexplained decreased urine output; or fever and graft tenderness and the episode was a case of biopsy proven AR (AR of Banff histopathologic classification Grade IA or higher as assessed by the blinded central pathologist); b: the reason for clinical suspicion was reported to be something other than: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; or an unexplained decreased urine output; or fever and graft tenderness; the episode was a case of biopsy proven AR, and the participant was treated for this episode. Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. AR is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection.
Time Frame: At 6 and 12 months post randomization
Population: ITT population: All randomized participants were summarized. N=number analyzed for Months 6 and 12
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 84 | 89
participants
  Total Number by Month 6 | 6 | 0
  By Month 6 Mild Acute (IA) | 1 | 0
  Month 6 Mild Acute (IB) | 1 | 0
  Month 6 Moderate Acute (IIA) | 3 | 0
  Month 6 Moderate Acute (IIB) | 1 | 0
  Month 6 Severe Acute (III) | 0 | 0
  Total Number by Month 12 | 6 | 0
  Month 12 Mild Acute (IA) | 1 | 0
  Month 12 Mild Acute (IB) | 1 | 0
  Month12 Moderate Acute (IIA) | 3 | 0
  Month 12 Moderate Acute (IIB) | 1 | 0
  Month 12 Severe Acute (III) | 0 | 0
Statistical Analysis 1: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); At Month 6, difference in percentage of participants with acute rejection (number with acute rejection/number randomized) using exact method; Test type: Superiority or Other; Difference in Percentage = 7.1, 95% CI 2-sided [2.1 to 14.9]
Statistical Analysis 2: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); At Month 12, difference in percentage of participants with acute rejection using exact method; Test type: Superiority or Other; Difference in Percentage = 7.1, 95% CI 2-sided [2.1 to 14.9]

3. Secondary Outcome: Percentage of Participants Surviving With a Functioning Graft, Have Graft Loss or Death (Graft Loss, Death, Death With Functioning Graft) By Month 6 and Month 12 Post Randomization
Description: Graft loss was defined as either functional loss or physical loss. Functional loss was defined as a sustained level of serum creatinine (SCr) ≥ 6.0 mg/dL (530 μmol/L) for ≥ 4 weeks or administration of a maintenance dialysis regimen for at least 56 days or impairment of renal function to such a degree that the participant undergoes re-transplantation.
Time Frame: At 6 and 12 months post randomization
Population: All participants who were randomized were summarized.
Measure: Number; unit: percentage of participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 84 | 89
percentage of participants
  Month 6 Surviving with Functioning Graft | 100.0 | 98.9
  Month 6 Graft Loss or Death | 0.0 | 1.1
  Month 6 Graft Loss | 0.0 | 0.0
  Month 6 Death | 0.0 | 1.1
  Month 6 Death with Functioning Graft | 0.0 | 1.1
  Month 12 Surviving with Functioning Graft | 100.0 | 98.9
  Month 12 Graft Loss or Death | 0.0 | 1.1
  Month 12 Graft Loss | 0.0 | 0.0
  Month 12 Death | 0.0 | 1.1
  Month 12 Death with Functioning Graft | 0.0 | 1.1
Statistical Analysis 1: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Participants surviving with a functioning graft by Month 6: For 95% Confidence Interval (CI) of difference, exact method was used; Test type: Superiority or Other; Percent Difference = 1.1, 95% CI 2-sided [-3.3 to 6.1]
Statistical Analysis 2: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Participants surviving with a functioning graft by Month 12: For 95% CI of difference, exact method was used; Test type: Superiority or Other; Percent Difference = 1.1, 95% CI 2-sided [-3.3 to 6.1]

4. Secondary Outcome: Number of Participants Who Had Any Study Drug Dose Alteration by Month 12 Due to Any Reason - Randomized and Treated Participants
Description: Reasons for study drug dose modification included categories of decline in renal function (as determined by the investigator), treatment of acute rejection, and other reasons. More than 1 reason could be given for dose alteration.
Time Frame: Month 12
Population: Participants who were randomized and received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Calcineurin Inhibitor (CNI): Participants received a CNI-based immunosuppressive regimen, CsA and tacrolimus TAC. CsA was to be adjusted to maintain a range of trough concentrations of 100 - 250 ng/mL. TAC doses were to be adjusted to maintain a range of trough serum concentrations of 5 - 10 ng/mL. During the LT period, participants were allowed to switch to the belatacept arm. In October 2011 (Year 3), the CNI arm was discontinued. CNI participants were considered to have completed treatment (not discontinued) at that time, if they did not switch to the belatacept arm.
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 83 | 88
participants
  Number with Dose Alteration (Any Reason) | 15 | 62
  Decline in renal function | 0 | 4
  Treatment of Acute Rejection | 0 | 0
  Other | 15 | 61

5. Primary Outcome: Mean Change From Baseline in Calculated Glomerular Filtration Rate (GFR) With Imputed Values to 12 Months Post Randomization - All Randomized Participants (Intent-to-Treat Population)
Description: Calculated GFR assessment used the modification of diet in renal disease (MDRD) formula. GFR was measured as mL/min/1.73 m^2. For death or graft loss participants, calculated GFR (cGFR) value 10 was used, for other participants who had a post baseline cGFR value missing, but had baseline value and at least 2 post baseline values available, which were at least 120 days apart, linear regression model was used to impute the cGFR value. Baseline = value at screening. Randomization/First Dose was on Day 1.
Time Frame: Baseline to 12 months post randomization
Population: Intent-to-Treat (ITT) population: all randomized participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Groups:
- Calcineurin Inhibitor (CNI): Participants received a CNI-based immunosuppressive regimen, CsA and TAC. CsA was to be adjusted to maintain a range of trough concentrations of 100 - 250 ng/mL. TAC doses were to be adjusted to maintain a range of trough serum concentrations of 5 - 10 ng/mL. During the LT period, participants were allowed to switch to the belatacept arm. In October 2011 (Year 3), the CNI arm was discontinued. CNI participants were considered to have completed treatment (not discontinued) at that time, if they did not switch to the belatacept arm by Year 3.
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 82 | 87
mL/min/1.73 m^2 | 7.0 (11.99) | 2.1 (10.34)

6. Secondary Outcome: Percentage of Participants With a Composite Endpoint of Death, Graft Loss and Acute Rejection at Month 12
Description: Percentage=number with composite divided by number randomized. Graft loss was functional loss or physical loss. Functional loss = sustained level of serum creatinine (SCr) ≥ 6.0 mg/dL for ≥ 4 weeks or administration of a maintenance dialysis regimen for at least 56 days or impairment of renal function to such a degree that participant undergoes re-transplantation. AR: if either a or b: (a) the reason for clinical suspicion was reported to be an unexplained rise of serum creatinine ≥ 25% from baseline; or an unexplained decreased urine output; or fever and graft tenderness and the episode was a case of biopsy-proven AR (grade IA or higher as assessed by the blinded central pathologist); (b) the reason for clinical suspicion was reported to be something other than: an unexplained rise of serum creatinine ≥ 25% from baseline; or an unexplained decreased urine output; or fever and graft tenderness; the episode was a case of biopsy-proven AR, and the participant was treated for it.
Time Frame: 12 Months post randomization
Population: All participants who were randomized were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 84 | 89
percentage of participants | 7.1 [1.6 to 12.7] | 1.1 [0.0 to 6.1]
Statistical Analysis 1: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Test type: Superiority or Other; Difference = 6.0, 95% CI 2-sided [-0.1 to 13.8]

7. Secondary Outcome: Percentage of Participants With New Onset Diabetes Mellitus - All Randomized Participants
Description: A participant who did not have diabetes prior to randomization is determined to have new onset diabetes mellitus if they received an antidiabetic medication for a duration of at least 30 days or at least two fasting plasma glucose (FPG) tests indicated that FPG is >=126 mg/dL. Percentage was the number of participants with new onset of diabetes mellitus divided by the number of participants without pre-randomization diabetes.
Time Frame: Month 12 post randomization
Population: Participants without pre-randomization diabetes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 59 | 68
percentage of participants | 1.7 [0.0 to 9.1] | 2.9 [0.4 to 10.2]

8. Secondary Outcome: Number of Participants With Anti-Donor Human Leukocyte Antigen (HLA) Positive Antibodies
Description: Samples were obtained at Day 1 (first dose), Week 24, and Week 52 (or end of therapy). This was a cumulative summary in that once a participant was positive, that participant remained positive for later time points. Evaluation of anti-donor HLA antibodies was performed by an external laboratory (Emory University, Atlanta, Georgia).
Time Frame: Month 6 and Month 12 Post Randomization
Population: Participants who had at least one test result or finding were summarized. n=number of participants analyzed at each specific time point.
Measure: Number; unit: participants
Groups:
- Belatacept 5 mg/kg: Belatacept 5 mg/kg given IV every 28 days.
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 82 | 83
participants
  Baseline (n=80,82) | 3 | 3
  Month 6 (n=82,82 | 3 | 4
  Month 12 (n=82, 83) | 3 | 4

9. Secondary Outcome: Mean Change From Baseline to Month 6 and to Month 12 in Serum Creatinine - All Randomized Participants
Description: Baseline was value at screening or prior to first dose of study drug. Serum creatinine was measured in milligrams per deciliter (mg/dL). Baseline = value at screening.
Time Frame: Baseline to Month 6 and Month 12 Post Randomization
Population: All randomized participants with baseline and laboratory value at specific time point were summarized.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 86
mg/dL
  Month 6 (n=81,82) | -0.1 (0.26) | -0.0 (0.20)
  Month 12 (n=81,86) | -0.1 (0.28) | -0.0 (0.21)

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Deaths, and Discontinuation Due to Adverse Events (AEs) From First Dose up to Month 12
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: First Dose (Day 1) to Month 12
Population: All randomized participants who received at least 1 dose of study drug were summarized.
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 83 | 88
participants
  Deaths | 0 | 1
  SAEs | 20 | 17
  Treatment Related SAEs | 9 | 4
  Discontinued due to SAEs | 1 | 0
  Treatment Related AEs | 24 | 27
  Discontinued due to AEs | 1 | 0

11. Secondary Outcome: Mean Change From Baseline in SF-36 Questionnaire Physical Component Score and in Mental Component Score at Month 12 - All Randomized Participants
Description: SF-36 was a Participant-Reported Quality of Life (QoL) Short Form (SF) questionnaire. The subscale in the mental component (MCS) part of the instrument ranged from 1 to 6 with 1=all of the time and 6= none of the time. The subscale for physical component (PCS) ranged from 1 to 3 with 1=Yes, limited a lot and 3=No, not limited at all. The subscale for the extent that physical health or emotional problems interfered with normal activities ranged from 1 to 5 with 1=not at all and 5= extremely. Baseline was at randomization or prior to first dose. Baseline = value at screening. The subscale scores were transformed using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life.
Time Frame: Baseline, Month 12
Population: All randomized participants who completed the questionnaire at baseline and at Month 12.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 64 | 75
units on a scale
  MCS (n=64, 75) | 0.3 (1.032) | -0.7 (0.959)
  PCS (n=64, 75) | 0.5 (0.808) | 0.8 (0.752)
Statistical Analysis 1: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Mental Component Scales (MCS); Test type: Superiority or Other; p = 0.4491, ANCOVA; Mean Difference (Net) = 1.1, 95% CI 2-sided [-1.7 to 3.9]
Statistical Analysis 2: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Physical Component Scales (PCS); Test type: Superiority or Other; p = 0.7892, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.5 to 1.9]

12. Secondary Outcome: Mean Change From Baseline to Month 12 for Eight Domain Scores of Quality of Life (QoL) Instrument SF-36 - All Randomized Participants
Description: SF-36 was a Participant-Reported Quality of Life (QoL) Short Form (SF) questionnaire measuring health-related quality of life (HRQL) covering 8 domains of physical and mental component summaries: physical function, role limitations due to physical problems, pain, general health perception, and vitality, social function, role limitations due to emotional problems, and mental health.
  All domains were scored using norm-based methods that standardized the scores to a mean of 50 and a standard deviation of 10 in the general population. The scores range from a minimum of 0 to a maximum of 100, with a higher score indicating better quality of life.
Time Frame: Baseline (screening) to Month 12
Population: Randomized participants with available questionnaires were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 75 | 79
units on a scale
  Bodily Pain (n=74,79) | 0.7 (0.979) | 0.3 (0.950)
  General Health (n=75,79) | 1.6 (0.921) | 0.9 (0.900)
  Mental Health (n=73,79) | 0.7 (0.913) | -0.1 (0.881)
  Physical Functioning (n=67,75) | -0.5 (0.840) | 0.8 (0.800)
  Role Emotional (n=75,79) | -1.4 (1.043) | -0.4 (1.021)
  Role Physical (n=75,79) | 0.5 (0.961) | 0.2 (0.939)
  Social Functioning (n=75,79) | 0.9 (0.929) | -0.5 (0.906)
  Vitality (n=73,79) | 0.2 (0.973) | -0.2 (0.940)

13. Secondary Outcome: Ridit Score at Month 12 - All Randomized Participants
Description: The Modified Transplant Symptom Occurrence and Symptom Distress Scale (MTSOSD-59R) was used to assess the occurrence (never, occasionally, regularly, almost always, always) and distress (0=no distress to 4=terrible distress) of symptoms associated with immunosuppressive therapies. Ridit (relative to an identified distribution) analysis (Fleiss JL. Statistical methods for rates and proportions. New York: John Wiley & Sons, Inc. 1991) was used. Ridit scores were calculated at 12 months for overall symptom occurrence score and overall symptom distress. The Ridit score reflects the probability that a score observed for an individual randomly selected from a group would be higher (worse symptom) than a score observed for a randomly selected individual from the reference group. The reference group was constituted by the frequency distribution of the responses of all participants on all items at baseline. The ridit of the reference group is by definition, 0.5.
Time Frame: Month 12
Population: All randomized participants with MTSOSD-59R data were analyzed.
Measure: Number; unit: Ridit score
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 46 | 45
Ridit score
  Symptom Distress (n=46,44) | 0.5162 | 0.5014
  Symptom Occurrence (n=46,45) | 0.5074 | 0.4998
Statistical Analysis 1: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Difference in Symptom Occurrence between treatment groups; Test type: Superiority or Other; Estimated Difference = .0076, 95% CI 2-sided [-.010 to .0252]
Statistical Analysis 2: Comparison: Belatacept 5 mg/kg vs Calcineurin Inhibitor (CNI); Difference in Symptom Distress between treatment groups; Test type: Superiority or Other; Estimated Difference = .0148, 95% CI 2-sided [-.002 to .0321]

14. Secondary Outcome: Number of Participants Meeting Marked Laboratory Abnormality Criteria From Baseline up to Month 12 - Randomized and Treated Participants
Description: Upper limits of normal (ULL). Leukocytes: < 2.0*10^3 cells per microliter (c/µL); Lymphocytes (absolute): < 0.5*10^3 c/µL; bilirubin: > 3.0*ULN milligrams per deciliter (mg/dL); Potassium: < 3.0 milliequivalents per liter (meq/L) or > 6.0 meq/L; Magnesium >2.6 meq/L; Sodium: < 130 meq/L; Phosphorus: < 2.0 mg/dL; Uric Acid: > 10 mg/dL. Baseline = value at screening.
Time Frame: Baseline up to Month 12
Population: All randomized participants who received at least one dose of study drug and had a laboratory value available post randomization. N= number of participants analyzed in all categories
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 83 | 87
participants
  Leukocytes Low | 0 | 1
  Lymphocytes Low | 4 | 0
  Bilirubin High | 0 | 1
  Potassium Low | 1 | 1
  Potassium High | 1 | 0
  Magnesium High | 5 | 1
  Sodium Low | 1 | 1
  Phosphorus Inorganic Low | 5 | 2
  Uric Acid High | 4 | 6

15. Secondary Outcome: Long Term Period: Mean Change From Baseline to 54 Months Post Randomization in Calculated GFR on Imputed Values at Specified Timepoints - Intent to Treat (ITT) Participants Who Entered LT Period
Description: ITT=participants randomized to their original treatment arm and who entered the LT period are presented. Baseline=value at screening. Calculated GFR assessment used the MDRD formula. GFR was measured as mL/min/1.73 m^2. For death or graft loss participants, calculated GFR (cGFR) value of 0 was imputed and carried forward after death or graft loss up to the end of the analysis period. Sponsor discontinued the CNI treatment arm in Year 3, and participants treated with CNI could elect to switch to belatacept. If a participant did not switch to belatacept, they were required to discontinue from the study. Therefore, efficacy results from Month 36 through Month 54 are difficult to interpret. No formal comparisons were planned between the belatacept and CNI treatment groups post Month 36, and the data up to the final database lock should be interpreted with caution.
Time Frame: Baseline, Month 3, 6, 12, 18, 24, 30, 36, 42, 48, 54
Population: Participants randomized to their original treatment arm who entered the LT Period (ITT - LT) and had data at baseline and at specific timepoints . Participants were grouped according to the treatment to which they were randomized (belatacept or CNI).
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
mL/min/1.73 m^2
  Month 3 (n=81, 81) | 5.1 (10.16) | 0.4 (9.92)
  Month 6 (n=80, 77) | 7.1 (11.94) | 2.3 (8.95)
  Month 12 (n=81, 81) | 7.1 (12.02) | 2.8 (9.70)
  Month 18 (n=81, 75) | 8.8 (13.88) | 0.1 (12.47)
  Month 24 (n=81, 78) | 8.8 (13.77) | -0.0 (14.84)
  Month 30 (n=80, 69) | 9.1 (16.10) | 0.1 (14.45)
  Month 36 (n=57, 52) | 7.7 (15.91) | 3.9 (17.46)
  Month 42 (n=71, 54) | 9.1 (17.56) | 0.6 (17.04)
  Month 48 (n=16, 32) | -1.7 (32.15) | 4.2 (18.03)
  Month 54 (n=14, 26) | -0.9 (35.69) | 2.4 (18.72)

16. Secondary Outcome: Long Term Period: Number of Participants With Acute Rejection (AR) - All Randomized Participants in LT Period
Description: AR was defined: if either a or b was satisfied: (a) the reason for clinical suspicion was reported to be an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; or an unexplained decreased urine output; or fever and graft tenderness and the episode was a case of biopsy proven AR (AR of Banff histopathologic classification grade IA or higher as assessed by the blinded central pathologist); (b) the reason for clinical suspicion was reported to be something other than: an unexplained rise of serum creatinine ≥ 25% from baseline creatinine; or an unexplained decreased urine output; or fever and graft tenderness; the episode was a case of biopsy proven AR, and the participant was treated for this episode. Banff 97 working classification of kidney transplant pathology was used to categorize the severity of the AR.
Time Frame: Post Month 12 up to Year 6 of the Study
Population: Participants, randomized to their original treatment arm, who entered the LT Period (ITT - LT) were analyzed. Participants were grouped according to the treatment to which they were randomized (belatacept or CNI).
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
participants
  Total Number | 5 | 4
  Mild Acute IA | 0 | 0
  Mild Acute IB | 1 | 1
  Moderate Acute IIA | 3 | 2
  Moderate Acute IIB | 1 | 1
  Severe Acute III | 0 | 0

17. Secondary Outcome: Long Term Period: Number of Participants Who Survived With a Functioning Graft or Survived With Pure Graft Loss or Death With Functioning Graft - ITT Participants Who Entered the LT Period
Description: Graft loss = either pure graft loss (participant survived to the end of the study period after graft loss) or death with functioning graft. Pure graft loss = either functional loss or physical loss. Functional loss = a sustained level of serum creatinine (SCr) ≥ 6.0 mg/dL (530 μmol/L) for ≥ 4 weeks or administration of a maintenance dialysis regimen for at least 56 days or impairment of renal function to such a degree that the participant undergoes re-transplantation. The table was designed with built-in redundancy to capture all possible combinations of death and/or graft loss, but not all lines can be summed to reach the total number surviving and the total number who die and/or lose grafts. If a participant experiences pure graft loss and dies at a later date independent of the graft loss event, they are counted only once in the cumulative tabulation of death or graft loss. Only the first event experienced by the participant counted toward the cumulative total.
Time Frame: Post Months 24, 36, 48, up to Year 6 of the Study
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
participants
  Month 24 Surviving with Functioning Graft | 80 | 80
  Month 24 Graft Loss or Death | 1 | 1
  Month 24 Graft Loss | 1 | 1
  Month 24 Death | 0 | 0
  Month 36 Surviving with Functioning Graft | 79 | 80
  Month 36 Graft Loss or Death | 2 | 1
  Month 36 Graft Loss | 1 | 1
  Month 36 Death | 1 | 0
  Month 36 Death with Functioning Graft | 1 | 0
  Month 48 Surviving with Functioning Graft | 78 | 80
  Month 48 Graft Loss or Death | 3 | 1
  Month 48 Graft Loss | 1 | 1
  Month 48 Death | 2 | 0
  Month 48 Death with Functioning Graft | 2 | 0
  up to year 6 Surviving with Functioning Graft | 76 | 80
  up to year 6 Graft Loss or Death | 5 | 1
  up to year 6 Graft Loss | 1 | 1
  up to year 6, Death | 4 | 0
  up to year 6 Death with Functioning Graft | 4 | 0

18. Secondary Outcome: Long Term Period: Percentage of Participants With New Onset Diabetes Mellitus Up to Month 36- All Randomized Participants Who Entered LT Period
Description: as for outcome 7
Time Frame: Baseline (screening) up to Month 36 post randomization
Population: Participants without pre-randomization diabetes, who were randomized and entered LT Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 58 | 62
percentage of participants | 6.9 [1.9 to 16.7] | 4.8 [1.0 to 13.5]

19. Secondary Outcome: Long Term Period: Number of Participants With SAEs, Death, Discontinuation Due to AEs - All Randomized Participants Who Entered the Long Term Period
Description: as for outcome 10
Time Frame: First dose after randomization (Day 1) to 56 days post last dose, up to Year 6 of the Study
Population: All participants who received at least 1 dose of study drug, were randomized to their original treatment arm, and who entered the LT Period (ITT - LT) were analyzed. Participants were grouped according to the treatment to which they were randomized (belatacept or CNI).
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
participants
  Deaths | 4 | 0
  SAEs | 45 | 40
  Treatment Related SAEs | 18 | 14
  Discontinued Due to SAEs | 1 | 2
  Treatment Related AEs | 38 | 43
  Discontinued Due to AEs | 1 | 3

20. Secondary Outcome: Long Term Period: Number of Participants With AEs of Special Interest - All Randomized Participants Who Entered the Long Term Period
Description: Prospectively identified events of special interest which were a subset of all AEs, and were either SAEs or non-serious AEs, included the following categories: Serious Infections, Thrombolic/embolic events, Autoimmune Disease, Malignancy, Peri-infusional reactions (only belatacept treatment group was IV) , Acute Peri-infusional events occurring within 24 hours of injection, Pulmonary Edema and Congestive Heart Failure. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose after randomization (Day 1) to last dose, plus 56 days, up to Year 6 of the Study
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
participants
  Malignancies | 8 | 9
  Serious Infections | 26 | 26
  Thrombolic/embolic | 3 | 0
  Peri-infusional Events | 37 | 0
  Acute Peri-infusional Events | 5 | 0
  Autoimmune Disease | 2 | 1
  Pulmonary Edema/Congestive Heart Failure | 3 | 2

21. Secondary Outcome: Long Term Period: Mean Change From Baseline to Month 54 in Serum Creatinine- ITT Participants Who Entered LT Period
Description: Baseline was value at screening. Serum creatinine was measured in mg/dL. Only participants who entered into Long Term Period were included in the analysis.
Time Frame: Baseline, Months 3, 6, 12, 18, 24, 30, 36, 42, 48, 54
Population: All participants who received at least 1 dose of study drug, were randomized to their original treatment arm, who entered the LT Period (ITT - LT), and had laboratory values were analyzed. Participants were grouped according to the treatment to which they were randomized (belatacept or CNI). n=entered LT Period with laboratory value available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
mg/dL
  Month 3 (n=81,81) | -0.1 (0.24) | 0.0 (0.21)
  Month 6 (n=81,77) | -0.1 (0.26) | -0.0 (0.19)
  Month 12 (n=81,81) | -0.1 (0.28) | -0.0 (0.21)
  Month 18 (n=80,75) | -0.1 (0.31) | 0.1 (0.77)
  Month 24 (n=80,77) | -0.1 (0.28) | 0.0 (0.37)
  Month 30 (n=78, 68) | -0.2 (0.35) | 0.0 (0.32)
  Month 36 (n=55, 51) | -0.1 (0.29) | -0.0 (0.39)
  Month 42 (n=68, 53) | -0.2 (0.30) | 0.0 (0.41)
  Month 48 (n=12, 31) | -0.2 (0.16) | -0.1 (0.30)
  Month 54 (n=10, 25) | -0.3 (0.25) | -0.1 (0.29)

22. Secondary Outcome: Long Term Period: Number of Participants Meeting Marked Laboratory Abnormality Criteria - All ITT Participants Who Entered the Long Term Period
Description: Upper limits of normal (ULN). Hemoglobin: < 8 g/dL; Platelet count: < 50*10^9 c/L; Leukocytes: < 2.0*10^3 c/µL; Lymphocytes (absolute): < 0.5*10^3 c/µL; Neutrophils: < 1.0*10^3 c/µL; Alanine Aminotransferase (ALT): > 5.0*ULN Units per liter (U/L); bilirubin: > 3.0*ULN mg/dL; Creatinine: > 3.0*ULN mg/dL; Calcium: < 7 mg/dL; Bicarbonate: > 12.5 mg/dL; Potassium: < 3.0 meq/L or > 6.0 meq/L; Magnesium >2.6 meq/L; Sodium: < 130 meq/L; Phosphorus: < 2.0 mg/dL; Uric Acid: > 10 mg/dL.
Time Frame: Baseline (Screening), up to Year 6 of the Study
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 81 | 81
participants
  Hemoglobin Low | 1 | 0
  Platelet Count Low | 1 | 1
  Leukocytes Low | 0 | 1
  Lymphocytes Low | 5 | 5
  Neutrophils Low | 1 | 2
  ALT High | 0 | 1
  Bilirubin High | 0 | 1
  Creatinine High | 0 | 1
  Calcium Low | 0 | 2
  Bicarbonate Low | 0 | 1
  Potassium Low | 2 | 1
  Potassium High | 1 | 3
  Magnesium High | 6 | 1
  Sodium Low | 2 | 1
  Phosphorus Inorganic Low | 7 | 3
  Uric Acid High | 7 | 7

23. Secondary Outcome: Long Term Period: Mean Change From Baseline to Month 54 in Systolic Blood Pressure
Description: Blood pressure was measured while the participant was sitting quietly for 5 minutes and was measured in millimeters of mercury (mmHg). Baseline was value at screening. Only those participants who entered long term period were evaluated.
Time Frame: Baseline, Months 6, 12, 18, 24, 30, 36, 42, 48, 54
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 80 | 78
mmHg
  Month 6 (n=78,73) | -3.6 (19.06) | -0.4 (17.52)
  Month 12 (n=77,71) | -4.6 (18.33) | -4.2 (16.26)
  Month 18 (n=77,1) | -4.4 (17.40) | 9.0 (NA) — Only 1 participant was available for analysis so standard deviation was not calculated.
  Month 24 (n=77,1) | -6.0 (17.94) | 4.0 (NA) — Only 1 participant was available for analysis so standard deviation was not calculated.
  Month 30 (n=75, 6) | -3.6 (17.94) | -0.5 (20.78)
  Month 36 (n=75,13) | -6.6 (17.49) | 1.2 (13.61)
  Month 42 (n=74, 29) | -5.4 (17.08) | -3.5 (19.33)
  Month 48 (n=73,32) | -4.4 (16.16) | -3.7 (14.35)
  Month 54 (n=72,33) | -4.9 (16.90) | -3.8 (12.96)

24. Secondary Outcome: Long Term Period: Mean Change From Baseline to Month 54 in Diastolic Blood Pressure
Description: Blood pressure was measured while the participant was sitting quietly for 5 minutes and was measured in mmHg. Baseline was value at screening. Only those participants who entered long term period were evaluated.
Time Frame: Baseline, Months 6, 12, 18, 24, 30, 36, 42, 48, 54
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI)
Number analyzed (Participants) | 80 | 78
mmHg
  Month 6 (n=78,73) | -2.0 (10.78) | -2.2 (10.50)
  Month 12 (n=77,71) | -2.5 (11.54) | -1.0 (11.04)
  Month 18 (n=77,1) | -1.7 (11.79) | 10.0 (NA) — Only 1 participant was available for analysis so standard deviation was not calculated.
  Month 24 (n=77,1) | -3.9 (10.19) | 13.0 (NA) — Only 1 participant was available for analysis so standard deviation was not calculated.
  Month 30 (n=75,6) | -1.8 (10.97) | 5.7 (9.14)
  Month 36 (n=75,13) | -1.9 (10.86) | -1.6 (7.69)
  Month 42 (n=74,29) | -1.7 (11.70) | -3.8 (10.99)
  Month 48 (n=73, 32) | -3.2 (10.53) | -3.6 (11.92)
  Month 54 (n=72, 33) | -1.1 (10.86) | -3.6 (11.72)

25. Secondary Outcome: Participants Who Switched From CNI to Belatacept in Long Term Period : Mean Change in Calculated GFR Based on Imputed Values From Day of Switch to Week 96 Post Switch
Description: Calculated GFR assessment used the MDRD formula. GFR was measured as mL/min/1.73 m^2. For death or graft loss participants, calculated GFR (cGFR) value 10 was used, for other participants who had a post baseline cGFR value missing, but had baseline value and at least 2 post baseline values available, which were at least 120 days apart, linear regression model was used to impute the cGFR value. Day of Switch = the first belatacept infusion day.
Time Frame: Day of Switch (first belatacept dose) to Week 96 Post Switch
Population: All randomized and treated participants who switched from CNI to belatacept during the long-term period were summarized. n=number of participants with data available at specific time point
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Groups:
- Belatacept 5 mg/kg in Participants Switched During LT Period: During the long term treatment period participants who had been randomized to CNI were allowed to switch to belatacept. For those switching to belatacept, the CNI dose was tapered and discontinued, after which they received belatacept 5 mg/kg IV every 2 weeks for 2 months. Thereafter, they received belatacept 5 mg/kg IV every 28 days.
Arm/Group | Belatacept 5 mg/kg in Participants Switched During LT Period
Number analyzed (Participants) | 38
mL/min/1.73 m^2
  Week 4 Post Switch (n=30) | 1.3 (5.85)
  Week 12 Post Switch (n=33) | 3.3 (9.88)
  Week 24 Post Switch (n= 29) | 2.1 (10.66)
  Week 48 Post Switch (n= 12) | 0.3 (7.75)
  Week 96 Post Switch (n= 8) | 0.1 (10.33)

26. Secondary Outcome: Participants Who Switched to Belatacept in Long Term Period: Number of Participants With AEs and SAEs
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Day of Switch = the first belatacept infusion day.
Time Frame: Day of Switch (first dose of belatacept ) to last dose plus 56 days, up to Year 6 of the Study
Population: All randomized and treated participants who switched from CNI to belatacept during the long-term period were summarized.
Measure: Number; unit: participants
Groups:
- Belatacept 5 mg/kg in Participants Switched During LT Period: During the long term treatment period participants were allowed to switch from CNI to belatacept. For those switching to belatacept, the CNI dose was tapered and discontinued, after which they received belatacept 5 mg/kg IV every 2 weeks for 2 months. Thereafter, they received belatacept 5 mg/kg IV every 28 days.
Arm/Group | Belatacept 5 mg/kg in Participants Switched During LT Period
Number analyzed (Participants) | 38
participants
  AEs | 32
  SAEs | 9

ADVERSE EVENTS:
Time Frame: Date of first dose to 56 days post final dose, up to June 2013 (approximately 80 months)
Description: Study initiated: January 2007; Study Completion: June 2013
Groups:
- Belatacept 5 mg/kg: Belatacept 5 milligrams per kilogram of body weight (mg/kg) given intravenously (IV) every 28 days. Adverse events reported for participants who were treated with only Belatacept throughout the study.
- Calcineurin Inhibitor (CNI): Participants received a calcineurin inhibitor (CNI)-based immunosuppressive regimen, Cyclosporin A (CsA) and tacrolimus (TAC). CsA was to be adjusted to maintain a range of trough serum concentrations of 100 - 250 nanograms per milliliter (ng/mL). TAC doses were to be adjusted to maintain a range of trough serum concentrations of 5 - 10 ng/mL. During the long term (LT) treatment period participants were allowed to switch to Belatacept treatment arm. In October 2011 (Year 3), the CNI arm was discontinued. CNI participants were considered to have completed treatment (not discontinued) at that time, if they did not switch to the Belatacept arm. Adverse events reported for participants who were treated with only CNI for the entire study and those who were later switched from Calcineurin Inhibitor (CNI) treatment to Belatacept 5 mg/kg during the LT period prior to their first Belatacept dose.
- Belatacept 5 mg/kg in Participants Switched During LT Period: During the long term treatment period participants were allowed to switch from CNI to Belatacept. For those switching to Belatacept, the CNI dose was tapered and discontinued, after which they received Belatacept 5 mg/kg IV every 2 weeks for 2 months. Thereafter, they received Belatacept 5 mg/kg IV every 28 days. Adverse events reported for participants who were switched from Calcineurin Inhibitor (CNI) treatment to Belatacept 5 mg/kg during the LT period on or after their first Belatacept dose.
Arm/Group | Belatacept 5 mg/kg | Calcineurin Inhibitor (CNI) | Belatacept 5 mg/kg in Participants Switched During LT Period
Serious Adverse Events (participants affected / at risk) | 45/83 | 40/88 | 9/38
Other Adverse Events (participants affected / at risk) | 78/83 | 74/88 | 27/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept 5 mg/kg (N=83) | Calcineurin Inhibitor (CNI) (N=88) | Belatacept 5 mg/kg in Participants Switched During LT Period (N=38)
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 3 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 0
Brain abscess (Infections and infestations) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nail bed infection (Infections and infestations) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 0
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0
Central nervous system infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hepatic cyst infection (Infections and infestations) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 2 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cystic lymphangioma (Congenital, familial and genetic disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2 | 0
Papilloma viral infection (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 2 | 0
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 1 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Necrotising retinitis (Eye disorders) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept 5 mg/kg (N=83) | Calcineurin Inhibitor (CNI) (N=88) | Belatacept 5 mg/kg in Participants Switched During LT Period (N=38)
Abdominal distension (Gastrointestinal disorders) | 5 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 7 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 9 | 7 | 1
Flatulence (Gastrointestinal disorders) | 5 | 0 | 0
Gastritis (Gastrointestinal disorders) | 6 | 7 | 0
Haematuria (Renal and urinary disorders) | 5 | 3 | 0
Leukocyturia (Renal and urinary disorders) | 6 | 0 | 0
Nasopharyngitis (Infections and infestations) | 21 | 12 | 3
Wound (Injury, poisoning and procedural complications) | 7 | 1 | 0
Blood creatinine increased (Investigations) | 6 | 4 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 12 | 4 | 1
Insomnia (Psychiatric disorders) | 11 | 5 | 0
Iron deficiency (Metabolism and nutrition disorders) | 6 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 7 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0
Onychomycosis (Infections and infestations) | 8 | 3 | 1
Renal impairment (Renal and urinary disorders) | 3 | 3 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Tinea versicolour (Infections and infestations) | 6 | 1 | 1
Dysuria (Renal and urinary disorders) | 12 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5 | 0
Hypertension (Vascular disorders) | 19 | 7 | 4
Pain (General disorders) | 5 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 7 | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Sinusitis (Infections and infestations) | 6 | 3 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 11 | 3 | 2
Fatigue (General disorders) | 4 | 5 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 13 | 1
Influenza (Infections and infestations) | 11 | 10 | 6
Proteinuria (Renal and urinary disorders) | 7 | 1 | 1
Weight increased (Investigations) | 5 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 18 | 12 | 1
Asthenia (General disorders) | 9 | 4 | 0
Bronchitis (Infections and infestations) | 14 | 6 | 5
Cataract (Eye disorders) | 5 | 4 | 0
Constipation (Gastrointestinal disorders) | 5 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 17 | 3
Diarrhoea (Gastrointestinal disorders) | 36 | 25 | 5
Headache (Nervous system disorders) | 16 | 9 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 0 | 1
Pyrexia (General disorders) | 12 | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Rhinitis (Infections and infestations) | 5 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 3 | 2
Weight decreased (Investigations) | 5 | 1 | 0
Chest pain (General disorders) | 8 | 3 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 0
Ear infection (Infections and infestations) | 5 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 8 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7 | 3
Paraesthesia (Nervous system disorders) | 11 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 2
Tremor (Nervous system disorders) | 1 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 11 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 8 | 2
Anxiety (Psychiatric disorders) | 5 | 8 | 1
Cytomegalovirus viraemia (Infections and infestations) | 5 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 5 | 1
Gout (Metabolism and nutrition disorders) | 4 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 19 | 10 | 9
Vomiting (Gastrointestinal disorders) | 5 | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypotension (Vascular disorders) | 6 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 0
Oedema peripheral (General disorders) | 20 | 7 | 1
Pharyngitis (Infections and infestations) | 6 | 12 | 5
Respiratory tract infection (Infections and infestations) | 8 | 8 | 0

LIMITATIONS AND CAVEATS:
CNI arm discontinued Year 3, and those not switching treatment discontinued from study. No formal comparisons in calculated GFR were planned post Month 36, and these data up to the final database lock should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.